CLINICAL TRIAL: NCT01859052
Title: Diet and Migraine Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team was unable to effectively conduct the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Drs Barbara Peterlin, Director of Headache Research, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIH1K23NS078345-01
Record Dates: First submitted 2013-05-10; First posted 2013-05-21 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Migraine; Obesity
Keywords: migraine; obesity; low fat diet; low carbohydrate diet
MeSH Terms: conditions — Migraine Disorders; Obesity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Obese migraineurs (Other): Low carbohydrate diet
  Interventions: Other: Low carbohydrate diet; Other: Low calorie low fat diet
- low-fat diet (Other): Obese Migraineurs
  Interventions: Other: Low carbohydrate diet; Other: Low calorie low fat diet
- Controls (Other): Controls receiving AHA diet recommendations
  Interventions: Other: AHA diet recommendations

INTERVENTIONS:
Other: Low carbohydrate diet — Subjects will follow the Atkins for Life diet. They will be given the book and a study dietitian will guide them through the induction, ongoing weight loss, pre-maintenance, and lifetime maintenance phases.
  Arms: Obese migraineurs; low-fat diet
Other: Low calorie low fat diet — The diet will be a nutritionally balanced, hypocaloric diet with a deficit of 750 kcal/day as guided by TEE. The goal is to match the calorie deficit to the low-CHO diet
  Arms: Obese migraineurs; low-fat diet
Other: AHA diet recommendations — given information in accordance with the diet and lifestyle recommendations of the American Heart Association.
  Arms: Controls

SUMMARY:
The purpose of this study is to look at two different diets (a low carbohydrate diet and a low fat diet) for migraine prevention in overweight or obese persons with migraine. The overall aim is to test the theory that diet will improve migraine frequency and that such improvements will be associated with favorable changes in body weight, inflammation, and heart health.

DETAILED DESCRIPTION:
Obesity is a risk factor for migraine. Further, in the past decade multiple lines of research have substantiated the presence of migraine headaches as a risk factor for CVD (eg. stroke). Migraineurs have also been demonstrated to have abnormal insulin responses, higher lipids and endothelial dysfunction. Limited data suggests a low fat diet may be of benefit in reducing migraine frequency; no studies have examined the efficacy of a low carbohydrate (ie. low glycemic) diet for migraine prevention in adults.. None of these studies examined the effects and potential mechanisms of such diet programs on CV health, body composition, and the inflammatory cascade in migraineurs. This 3 -month study addresses the efficacy and potential mechanisms of two different diets, (a low carbohydrate diet and a low fat diet) for migraine prevention in a clinical cohort of overweight or obese persons with migraine. The overall aim is to test the hypothesis that each behavioral intervention will improve migraine frequency and that such improvements will be associated with favorable changes in body composition, inflammation, and CV parameters.

Hypothesis 1.1 The mean monthly migraine frequency will be decreased in those who maintain a low-fat diet or low-carbohydrate diet for 3 months as compared to controls.

Hypothesis 1.2 Participants randomized to the diets will demonstrate favorable changes in body composition (eg. decrease in adipose tissue volume on magnetic resonance imaging (MRI) and body fat on DEXA), inflammatory markers (eg. decrease in adipocytokine levels), and CV parameters (eg. improved cholesterol panel, glucose levels and markers of arterial stiffness) as compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (BMI between 25 and 42)
* women
* >18 years and < 50 years old
* Migraine meeting ICHD criteria for at least 6 months prior to screening
* headache frequency documented > 2 and < 10 headache days per month
* BP inclusion criteria are SBP <160 or DBP <100 mm Hg

Exclusion Criteria:

* hypocaloric diet (must be weight stable for prior 3 months)
* Self-report of alcohol or substance abuse in the past year or current treatment
* Type 1 or 2 diabetes

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mean change in headache frequency | 3 months.
  Change in headache frequency from baseline to 3 months
Mean change in body composition | 3 months
  The mean change in body composition from the baseline phase to 3 months
The mean change in inflammatory markers | 3 month
  The mean change in inflammatory markers from baseline to 3 months

SECONDARY OUTCOMES:
Proportion of patients responding to treatment | 3 months
  Proportion of participants responding to weight loss program as measured by a 21% or more reduction in mean monthly migraine frequency

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Peterlin, DO, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Johns Hopkins Bayview Headache Center, Baltimore, Maryland, United States